CLINICAL TRIAL: NCT02474381
Title: Efficacy Study of Autologous Endothelial Progenitor Cells Treatment of Diabetic Foot With Infrapopliteal Arterial Stenosis/Occlusion
Brief Title: Autologous Endothelial Progenitor Cells Treatment of Diabetic Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Maoquan Li, Chief of Interventional Department, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-xjs-06
Record Dates: First submitted 2015-06-10; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2012-12

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPCs plus PTA (Experimental): Intra-arterial infusion of autologous CD133+ cells on diabetic subjects with PAD,plus angioplasty
  Interventions: Biological: EPCs plus PTA
- Single PTA (Active Comparator): Angioplasty of arteries below tibial plateau level only
  Interventions: Device: Single PTA

INTERVENTIONS:
Biological: EPCs plus PTA — Intra-arterial infusion of autologous CD133+ cells on diabetic subjects with PAD,plus angioplasty
  Arms: EPCs plus PTA
Device: Single PTA — Angioplasty of arteries below tibial plateau level only
  Arms: Single PTA

SUMMARY:
The vascular pathologic basis of diabetic foot include arterial obstruction and micro-circulation defects.The latest technology of arterial reconstruction can only rebuild blood flow of anterior,posterior tibial artery and peroneal artery.Endothelial progenitor cells have been proved to integrate into damaged vascular endothelium and improve vasculogenesis in vitro and in animal experiment.Therefore endothelial progenitor cells are supposed to improve the micro-circulation status of diabetic foot patients.In this trial,the investigators recuit diabetic foot patients with infrapopliteal arterial obstructive disease,treat them with autologous endothelial progenitor cells after intraluminal intervention,and observe the therapeutic efficacy comparing to single intraluminal intervention.

DETAILED DESCRIPTION:
Study design The study was a prospective, non-random¬ized trial conducted at 2 centers in east China - Tenth People's Hospital of Tongji University and Nanjing First Hospital. The ethic committee at each center approved the protocol, and all patients provided written informed consent. All patients enrolled were assigned to CD133+ cells treatment group (CD133+ group) and control group of their own volition. This study is to evaluate the efficacy and immune-regulatory impact of intra-arterial infusion of autologous CD133+ cells on diabetic subjects with PAD.

Patient enrollment and grouping Diabetic PAD patients aged ≥18 years with Rutherford categories 2 to 5 were included to assess the eligibility for this study. All patients, who agreed to participate in the study, could voluntary choose whether or not to receive autologous CD133+ progenitor cell treatment.

In this study, CD133+cells were used to stimulate angiogenesis and reconstruct efficient microvascular blood supply, therefore similar hemodynamic status in main branch was essential to meet homogeneityin both groups before patient entry. The candidates, who failed for intraluminal revascularization of infra-aorta (iliac and femoral-popliteal)and 1 infra-popliteal (anterior/posterior tibial, fibular) arteries of the affected limb, would be excluded from the study.

Other exclusion criterion were as follows: ① Hemoglobin < 10 mg/dl, ② creatinine clearance < 30 ml/min, ③ previous history of stem/progenitor cell therapy, ④ paralysis because of central neural system disease, ⑤ accidental amputation or bone fracture of target limb because of trauma after entry, ⑥ stop of anti-platelet medication after entry, ⑦ smoking or re-smoking after entry, ⑧ malignant tumor.

Treatment of infra-aorta & infra-popliteal artery lesion Computed tomographic angiography (CTA) was performed to firstly analyze the condition of vascular lesion and then digital subtraction angiography (DSA) was performed to precisely identify the lesions of infra-aorta and the infra-popliteal arteries before treatment.

The treatment of infra-aorta artery lesion was restrictedly performed with intraluminal technique (balloon dilation and/or stent implantation) nevertheless the grade of the lesion according to TASC II classification. The arterial sheath was introduced into the contralateral femoral artery, and then the revascularization of the target limb was accomplished by antegrade approach.

After the previous procedure, the lesions of the infra-popliteal arteries were re-evaluated by DSA. By means of balloon dilation, at least one of the anterior/posterior tibial and fibular arteries achieved an obvious direct blood supply to the foot.

The goal of the above procedures is to completely restore the normal main trunk hemodynamic status of the target limb.

Autologous CD133+ cells collection and preparation After successful revascularization of infra-aorta and infra-popliteal procedure, 100ml peripheral blood was collected through the femoral artery sheath in patients and sent to East China Stem Cell Bank for CD133+ cells sorting and enrichment. Mononuclear cells are separated from the whole blood by density gradient centrifugation with Ficoll separating medium, then CD133+ cells are selected using magnetic-activated cell sorting. The selected cells were mixed with 50ml sodium chloride injection, which contains human albumin and heparin sodium in the blood bag, and then sent back to hospital stored in 4℃. All collection and preparing procedures were finished within 6 hours.

The selected cells also need to take a quality test, otherwise the cells would be discarded and the source patient would be excluded from the study. The quality standards are as following: cell number ≥ 1×107, no visible precipitate in cell suspension, viable cell ≥90%, endotoxin ≤ 2EU/ml Cell Infusion Procedure A catheter was introduced into the popliteal artery of the target limb at tibial plateau level. The CD133+ cells suspension was drawn into a 50ml syringe and infused through the catheter by an injection pump timing to 30 minutes.

For the control group, 50ml cell-free sodium chloride injection containing human albumin and heparin sodium were infused through the catheter as placebo.

Medication and life style change Both groups were asked to receive continuous medication for the diabetes, hyperlipidemia and hypertension under the advices of specialized physicians. Anti-platelet treatment with 100mg of enteric-coated aspirin and 75mg clopidogrel daily, as well as statins administration for stabilizing of the arterial plaque, was also demanded.

Besides these medications, all candidates were restrictedly asked to quit smoking after entry.

Follow-up and Endpoints The patients were followed up at 18 months. The primary endpoints were defined as the aggravation of ulcer (developing new or larger or deeper ulcers) and the amputation (above metatarsal level). The ulcer healing and amputation status were observed monthly.

The change of Rurtherford classification, TcPO2 of dorsum pedis and ABI were recorded to evaluate the blood perfusion of the limb at 6 and 18 month as the second endpoints.

As proven, the stem cells promote angiogenesis through stimulation of endothelial cell proliferation, migration, and survival by paracrine of high levels of vascular endothelial growth factor (VEGF) [9]. In addition to the regenerative properties, stem cells have an immune-regulatory capacity and induce immunosuppressive effects in a series of situations [10]. Human stem cells have been found to suppress Interleukin-6 (IL-6) expression in activated macrophages, which plays a key role in inflammatory response in wound healing [11]. Thus, the serum concentrations of VEGF and IL-6 before and at 1, 2, 4 week after the CD133+ cells infusion were tested to evaluate the pro-angiogensis and immunoregulatory impact of the procedure and its duration.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic PAD patients aged ≥18 years with Rutherford categories 2 to 5

Exclusion Criteria:

* Hemoglobin < 10 mg/dl
* Creatinine clearance < 30 ml/min
* Previous history of stem/progenitor cell therapy
* Paralysis because of central neural system disease
* Accidental amputation or bone fracture of target limb because of trauma after entry
* Stop of anti-platelet medication after entry
* Smoking or re-smoking after entry
* Malignant tumor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Infrapopliteal arterial patency of the affected extremity | Every 3 month until 1year after the treatment
  Ultrasonography deployed to assess the patency

SECONDARY OUTCOMES:
Amputation rate of the affected extremity | At 6 month and 1 year after the treatment
  Whether the affect extremity amputated

CONTACTS AND LOCATIONS:
Overall Officials: Chenhui Lu, Ph.D, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth people's hospital, Tongji university, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Wu T, Liu Y, Wang B, Li G. The roles of mesenchymal stem cells in tissue repair and disease modification. Curr Stem Cell Res Ther. 2014;9(5):424-31. doi: 10.2174/1574888x09666140616125446. PMID 24998241
- [Result] Invernici G, Emanueli C, Madeddu P, Cristini S, Gadau S, Benetti A, Ciusani E, Stassi G, Siragusa M, Nicosia R, Peschle C, Fascio U, Colombo A, Rizzuti T, Parati E, Alessandri G. Human fetal aorta contains vascular progenitor cells capable of inducing vasculogenesis, angiogenesis, and myogenesis in vitro and in a murine model of peripheral ischemia. Am J Pathol. 2007 Jun;170(6):1879-92. doi: 10.2353/ajpath.2007.060646. PMID 17525256